CLINICAL TRIAL: NCT01047371
Title: Why in Hospital - Factors Determining Time to Discharge Readiness After Arthroplasty Surgery: An Prospective Observational Study
Brief Title: Why in Hospital - Factors Determining Time to Discharge Readiness After Arthroplasty Surgery
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Lundbeck Foundation (Other)
Responsible Party: Principal Investigator, Troels Haxholdt Lunn, MD, Hvidovre University Hospital
Other Study IDs: 1234; 5678
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Pain; Nausea; Vomiting; Dizzyness; Fatigue; Organizational Concerns; Ect.
MeSH Terms: conditions — Pain; Nausea; Vomiting; Dizziness; Fatigue; Epilepsy, Rolandic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Osteoarthrosis: All consecutive patients scheduled for total hip or knee arthroplasty

SUMMARY:
The purpose of this study is to evaluate patient related factors determining length of stay in hospital after arthroplasty surgery.

DETAILED DESCRIPTION:
To evaluate why the patient is in hospital after surgery, when predefined discharge criteria are met, which patient related clinical problems hinder fulfilling of the discharge criteria, and to evaluate actual length of stay in hospital.

All consecutive patients scheduled for total hip or knee arthroplasty are included in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip or knee arthroplasty

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients scheduled for total hip or knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Patient related factors determining length of stay in hospital | Daily (average 2 days)

SECONDARY OUTCOMES:
Length of stay in hospital | At discharge (average 2 days)
Time till fulfilling of predefined discharge criteria | At discharge (average 2 days)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Husted, MD, Study Director — Hvidovre University Hospital; Troels H. Lunn, M.D, Principal Investigator — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark